CLINICAL TRIAL: NCT06307925
Title: A Phase I Open-label, Multi-center, Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics and Antitumor Activity of HC010 in Patients With Advanced Solid Tumors
Brief Title: A Phase I Study to Evaluate the Safety, Pharmacokinetics and Antitumor Activity of HC010 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC010-001
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tumor; Non-small cell lung cancer; Hepatocellular carcinoma; colorectal cancer; cervical cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Hepatocellular; Colorectal Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dose-escalation phase (Experimental): HC010 0.15mg/kg to 20mg/kg Q2w/28d intravenous infusion
  Interventions: Drug: HC010
- dose expansion phase (Experimental): Fixed dose of HC010 Q2w/28d intravenous infusion
  Interventions: Drug: HC010

INTERVENTIONS:
Drug: HC010 — HC010 Q2W/28d intravenous infusion

SUMMARY:
This clinical trial is a multicenter, open, single-arm, non-randomized, dose-escalation and dose-expansion, phase I clinical study in patients with advanced recurrent or metastatic solid tumors.The goal of this study is to evaluate the safety and tolerability of HC010 monotherapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This clinical trial is a multicenter, open, single-arm, non-randomized, dose-escalation and dose-expansion, phase I clinical study in patients with advanced recurrent or metastatic solid tumors.The goal of this study is to evaluate the safety and tolerability of HC010 monotherapy in patients with advanced solid tumors.Enrollment is for patients with advanced adult solid tumors (including but not limited to non-small cell lung cancer, hepatocellular carcinoma, colorectal cancer, cervical cancer, triple-negative breast cancer, gastric cancer/gastroesophageal junction adenocarcinoma, ovarian cancer, pancreatic cancer, bladder cancer, and renal cancer) who have either failed to respond to standard of care or who are unable to receive/do not have access to standard of care.Subjects received HC010 monotherapy by intravenous infusion every two weeks in 1 cycle of 28 days, and were treated until completion of 2 years of study treatment, disease progression, intolerable toxicity, withdrawal of informed consent, loss to follow-up, death, or fulfillment of other criteria for termination of treatment, whichever occurred first. The primary study endpoints were safety and tolerability, maximum tolerated dose (MTD) and/or recommended dose for phase II clinical studies (RP2D); secondary endpoint indicators included pharmacokinetic indicators, efficacy indicators [objective response rate (ORR), duration of response (DoR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS)], immunogenicity indicators such as anti-drug antibody (ADA) and neutralizing antibody (Nab). Exploratory endpoints included the pharmacokinetic (PD) index of HC010, the relationship between peripheral blood T-cell receptor occupancy (RO) and safety and efficacy, as well as the correlation between PD-L1 expression level in tumor tissues and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in this clinical trial, understanding and following the research protocol, and voluntarily signing the Informed Consent Form (ICF).
2. Age ≥18 and ≤75, male or female.
3. Participants with histologically or cytologically confirmed diagnosis of advanced solid tumors who have failed standard therapy or for whom no standard therapy is available.
4. Participants must have at least one measurable lesion according to RECIST Version1.1
5. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1
6. Hepatocellular carcinoma patients with Child-Pugh score ≤ 7
7. Expected survival time is at least 3 months
8. Adequate organ function: neutrophil count≥1.5×109/L,platelet count ≥100×109/L,hemoglobin≥90g/L,alanine aminotransferase and aspartate aminotransferase ≤2.5×upper limit of normal (ULN); patients with hepatocellular carcinoma or concomitant hepatic metastases ≤5.0×ULN, total bilirubin ≤1.5×ULN, renal function and cardiopulmonary function are basically normal.
9. Subjects should provide, whenever possible, freshly obtained or archived tumor tissue sample prior to study treatment that can be used for biomarker analysis
10. Participants of childbearing potential (males and females) must agree to effective contraception for at least 90 days from the time of signing the informed consent form to the time of the last dose; females of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose of the HC010

Exclusion Criteria:

1. Receipt of any interventional clinical trial treatment or other systemic chemotherapy, radiotherapy, etc. within 28 days or 5 half-lives (whichever is shorter) prior to the first dose of the HC010; Receipt of herbal or proprietary Chinese medicine with an anti-tumor indication within 2 weeks prior to the first dose of HC010;
2. Underwent surgery, experienced severe trauma, etc,within 4 weeks prior to the first administration of HC010 ;
3. Receipt of systemic glucocorticoids (prednisone >10 mg/day or equivalent doses of similar drugs) or other immunosuppressive agents within 2 weeks prior to the first dose of HC010;
4. Receipt of immunomodulatory drugs within 2 weeks prior to the first dose of HC010;
5. Receipt of live attenuated vaccination within 4 weeks prior to the first dose of HC010;
6. Patients who have received biomolecule therapy for anti-programmed death receptor 1 (PD-1)/programmed death ligand (PD-L1), anti-cytotoxic T-lymphocyte antigen 4 (CTLA-4), and anti-vascular endothelial growth factor (VEGF) targets in prior antitumor therapy;
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v5.0 Grade≤1;
8. History of immune-related adverse event (irAE) leading to permanent discontinuation from prior immunotherapy ,or grade ≥3 toxicity related to anti-angiogenic therapy from prior anti-angiogenic therapy；
9. Previous allogeneic hematopoietic stem cell transplantation or organ transplantation；
10. Patients with known active brain metastases, or the presence of meningeal metastases, spinal cord compression, or molluscum contagiosum disease；
11. Combination of other malignancies within 5 years prior to the first dose; excludes radically treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, papillary thyroid carcinoma and/or radically resected carcinoma in situ;
12. Patients with active autoimmune disease, or a history of autoimmune disease；
13. Infections: 1) active hepatitis B and C; Note: HBsAg and/or hepatitis B core antibody (HBcAb) positive individuals with HBV DNA ≥500 IU/ml (≥2000 IU/ml in patients with hepatocellular carcinoma) tested within 28 days prior to the initiation of treatment are eligible for inclusion.2) known history of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS); 3) known active syphilis; 4) active tuberculosis; 5) active infection within two weeks prior to first dose of HC010;
14. Unstable systemic disease, including but not limited to, severe cardiovascular disease; pleural effusion, pericardial effusion or peritoneal effusion requiring repeated drainage;
15. Severe bleeding tendencies or coagulation disorders;
16. History of non-infectious pneumonia/interstitial lung disease requiring systemic glucocorticoid therapy;
17. Females who are pregnant or breastfeeding;
18. Inappropriate for this study in the opinion of the investigator;
19. History of systemic hypersensitivity or anaphylaxis to any component of HC010.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-03-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity | 28 days
  Incidence of dose-limiting toxicity
Adverse events | 2 years
  Adverse events
serious adverse events | 2 years
  serious adverse events
Maximum Tolerated Dose | 2 years
  Maximum Tolerated Dose
Recommended Dose for Phase II Clinical Studies | 2 years
  Recommended Dose for Phase II Clinical Studies

SECONDARY OUTCOMES:
pharmacokinetics:Cmax | 2 years
  pharmacokinetics:Cmax
Objective response rate | 2 years
  Objective response rate (ORR)
duration of response | 2 years
  duration of response (DoR)
progression-free survival | 2 years
  progression-free survival
overall survival | 2 years
  overall survival
Disease control rate | 2 years
  Disease control rate
pharmacokinetics:AUC0-last | 2 years
  pharmacokinetics:AUC0-last
pharmacokinetics:tmax | 2 years
  pharmacokinetics:tmax
pharmacokinetics:Vd | 2 years
  pharmacokinetics:Vd

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No